CLINICAL TRIAL: NCT06945107
Title: A Phase III, Multicenter, Randomized, Double-Blind, Active-Controlled Study to Evaluate the Efficacy and Safety of Switching to Picankibart in Patients With Plaque Psoriasis With an Inadequate Response to Interleukin-17 Monoclonal Antibody Therapy
Brief Title: A Study of Switching to Picankibart in Chinese Patients With Plaque Psoriasis With an Inadequate Response to Interleukin-17 Monoclonal Antibody Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biopharmaceutical Technology (Hangzhou) Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI112A303CN
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — secukinumab; ixekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Picankibart treatment group (Experimental): The participants in this group will receive picankibart 200mg SC at Weeks 0, 4, 8, 20 and 32.
  Interventions: Drug: Picankibart; Drug: Placebo
- IL-17 mAb continued treatment group (Active Comparator): The participants in this group will receive the original IL-17 mAb at Weeks 0, 4, 8 and 12, followed by picankibart 200mg SC at Weeks 16, 20, 24 and 36.
  Interventions: Drug: Picankibart; Drug: Secukinumab; Drug: Placebo; Drug: Ixekizumab

INTERVENTIONS:
Drug: Picankibart — The participants in picankibart treatment group will receive picankibart 200mg SC at Weeks 0, 4, 8, 20 and 32.
  The participants in IL-17 mAb continued treatment group will receive picankibart 200mg SC at Weeks 16, 20, 24 and 36.
Drug: Secukinumab — The participants in IL-17 mAb continued treatment group who have received secukinumab before enrollment, will receive secukinumab 300mg SC at Weeks 0, 4, 8 and 12.
  Arms: IL-17 mAb continued treatment group
Drug: Placebo — The participants in picankibart treatment group will receive placebo SC at Weeks 12, 16, 24 and 36.
  The participants in IL-17 mAb continued treatment group will receive placebo SC at Week 32.
Drug: Ixekizumab — The participants in IL-17 mAb continued treatment group who have received ixekizumab before enrollment, will receive ixekizumab 80mg SC at Weeks 0, 4, 8 and 12.
  Arms: IL-17 mAb continued treatment group

SUMMARY:
This multicenter, randomized, double-blind, active-controlled study aims to evaluate the efficacy and safety of picankibart in Chinese patients with plaque psoriasis who demonstrated inadequate responses to interleukin-17 (IL-17) monoclonal antibody therapy and subsequently switched to picankibart. The trial will enroll approximate 310 participants with confirmed plaque psoriasis diagnosis and a poor response to IL-17 monoclonal antibody treatment. The study includes a 4-week screening phase, followed by an active treatment period of either 36 weeks, and concludes with a safety follow-up assessment at Week 48.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years and ≤75 years.
2. Diagnosed with plaque psoriasis for ≥6 months, with or without psoriatic arthritis.
3. Regular use of secukinumab or ixekizumab according to the label information for at least 16 weeks prior to baseline (actual dose received ≥80% of the standard dose per instructions during the 16 weeks before baseline), with sufficient documented rationale for medication use.
4. At both screening and baseline, meet the criteria of sPGA (Static Physician's Global Assessment) ≥2 and body surface area (BSA) involvement ≥3%, along with the investigator's assessment of inadequate response to the original IL-17 monoclonal antibody therapy, warranting a switch to biologic treatment.
5. Full understanding of the trial objectives, basic knowledge of the pharmacological effects and potential adverse reactions of the investigational product, and voluntary provision of written informed consent in accordance with the principles of the Helsinki Declaration.

Exclusion Criteria:

1. Diagnosed with guttate psoriasis, pustular psoriasis, or erythrodermic psoriasis during screening or at baseline;
2. Previous diagnosis of drug-induced psoriasis (e.g., psoriasis induced by beta blockers, calcium channel inhibitors, etc.);
3. Prior use of picankibart or IL-23 inhibitors;
4. Received two biological agents for psoriasis treatment within 16 weeks prior to screening;
5. Received topical treatments that may affect psoriasis evaluation within 2 weeks before the first administration of the investigational product (including but not limited to glucocorticoids, vitamin D3 derivatives, retinoids, calcineurin inhibitors, keratoplastics, and combination therapies);
6. Received conventional systemic medications that may affect psoriasis evaluation within 4 weeks before the first administration of the investigational product (including but not limited to methotrexate, cyclosporine, retinoids, azathioprine, leflunomide, mycophenolate mofetil, sulfasalazine, glucocorticoids, apremilast, JAK inhibitors such as tofacitinib/baricitinib/upadacitinib, TYK2 inhibitors such as deucravacitinib, or Chinese herbal medicines for psoriasis);
7. Use of natalizumab, or B-cell/T-cell modulators (e.g., rituximab, abatacept, visilizumab) within 12 months before the first administration of the investigational product;
8. Received phototherapy for psoriasis within 1 month before the first administration of the study drug, and/or unwillingness to avoid prolonged sun exposure and other UV light sources (e.g., sunbathing/tanning devices) during the study;
9. Received investigational biological agents within 6 months, any investigational therapy within 30 days, study drugs within 5 half-lives (whichever is longer), or current participation in clinical trials before the first administration of the investigational product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-06-07 (Estimated); Study Completion 2027-01-19 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants achieving static Physician's Global Assessment (sPGA) score of clear (0) or almost clear (1) | Week 16
  The static Physician's Global Assessment (sPGA) is a 5-point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. A lower score indicates less body coverage, with 0 being clear and 1 being almost clear.

SECONDARY OUTCOMES:
The percentage of participants achieving a Psoriasis Area and Severity Index (PASI) 75 response | Week 16
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 75 is defined as at least a 75% reduction in PASI score compared with the Baseline PASI score.
The percentage of participants achieving a PASI 90 response | Week 16
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score.
The percentage of participants achieving sPGA=0 | Week 16
  The static Physician's Global Assessment (sPGA) is a 5-point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. A lower score indicates less body coverage, with 0 being clear.
The percentage of participants with involved body surface area (BSA) <3% (or ≥75% reduction relative to baseline) | Week 16
  The area of involved body surface area (BSA) will be estimated by the Investigator as a percentage of the subject's total body surface area wherein the area of the subject's palm will be considered as 1% of total BSA. The involved BSA ranges from 0% to 100%, where a lower BSA indicates less involved skin.
The percentage of participants achieving sPGA=0/1 and with involved BSA <3% (or ≥75% reduction relative to baseline) | Week 16
  The static Physician's Global Assessment (sPGA) is a 5-point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. A lower score indicates less body coverage, with 0 being clear and 1 being almost clear. The area of involved involved body surface area (BSA) will be estimated by the Investigator as a percentage of the subject's total body surface area wherein the area of the subject's palm will be considered as 1% of total BSA. The involved BSA ranges from 0% to 100%, where a lower BSA indicates less involved skin.
The percentage of participants achieving Dermatology Life Quality Index (DLQI)=0/1 (for participants with baseline DLQI >1 only) | Week 16
  The Dermatology Life Quality Index (DLQI) is a self-administered, 10-question questionnaire covering 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and bother with psoriasis treatment). The response options range from 0, not affected at all, to 3, very much affected. This gives an overall range of 0 to 30 where lower scores mean better quality of life.
The percentage of participants achieving a PASI 100 response | Week 16
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 100 is defined as a 100% reduction in PASI score compared with the Baseline PASI score.
The change from baseline in PASI score | Week 16
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.
The change from baseline in involved BSA | Week 16
  The area of involved body surface area (BSA) will be estimated by the Investigator as a percentage of the subject's total body surface area wherein the area of the subject's palm will be considered as 1% of total BSA. The involved BSA ranges from 0% to 100%, where a lower BSA indicates less involved skin.
The percentage of participants achieving sPGA=0/1 | Week 44
  The static Physician's Global Assessment (sPGA) is a 5-point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. A lower score indicates less body coverage, with 0 being clear and 1 being almost clear.
The percentage of participants achieving sPGA=0 | Week 44
  The static Physician's Global Assessment (sPGA) is a 5-point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. A lower score indicates less body coverage, with 0 being clear.
The percentage of participants with involved BSA<3% (or ≥75% reduction relative to baseline) | Week 44
  The area of involved body surface area (BSA) will be estimated by the Investigator as a percentage of the subject's total body surface area wherein the area of the subject's palm will be considered as 1% of total BSA. The involved BSA ranges from 0% to 100%, where a lower BSA indicates less involved skin.
The percentage of participants achieving sPGA=0/1 and with involved BSA <3% (or ≥75% reduction relative to baseline) | Week 44
  The static Physician's Global Assessment (sPGA) is a 5-point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. A lower score indicates less body coverage, with 0 being clear and 1 being almost clear. The area of involved BSA will be estimated by the Investigator as a percentage of the subject's total body surface area wherein the area of the subject's palm will be considered as 1% of total BSA. The involved BSA ranges from 0% to 100%, where a lower BSA indicates less involved skin.
The percentage of participants achieving DLQI=0/1 (for participants with baseline DLQI >1 only) | Week 44
  The Dermatology Life Quality Index (DLQI) is a self-administered, 10-question questionnaire covering 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and bother with psoriasis treatment). The response options range from 0, not affected at all, to 3, very much affected. This gives an overall range of 0 to 30 where lower scores mean better quality of life.
The percentage of participants achieving a PASI 75 response | Week 44
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 75 is defined as at least a 75% reduction in PASI score compared with the Baseline PASI score.
The percentage of participants achieving a PASI 90 response | Week 44
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score.
The percentage of participants achieving a PASI 100 response | Week 44
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 100 is defined as a 100% reduction in PASI score compared with the Baseline PASI score.
The change from baseline in PASI score | Week 44
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.
The change from baseline in involved BSA | Week 44
  The area of involved body surface area (BSA) will be estimated by the Investigator as a percentage of the subject's total body surface area wherein the area of the subject's palm will be considered as 1% of total BSA. The involved BSA ranges from 0% to 100%, where a lower BSA indicates less involved skin.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Hospital of Shandong First Medical University (Shandong Provincial Hospitial of Dermatology), Jinan, Shandong, China